CLINICAL TRIAL: NCT01793649
Title: A Phase 1, Randomized, Double-Blind, Cross-Over, Vehicle-Controlled, Single-Dose Study To Characterize The Effect of GS-5737 Enhancement of Mucociliary Clearance (MCC) In Healthy Subjects
Brief Title: A Phase 1 Study to Characterize the Effect of GS-5737 Enhancement of Mucociliary Clearance (MCC) in Healthy Subjects
Status: Terminated | Phase: Phase 1 | Type: Interventional
Sponsor: Gilead Sciences (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Treatment
Other Study IDs: GS-US-234-0103
Record Dates: First submitted 2013-02-14; First posted 2013-02-15 (Estimated); Last update posted 2014-03-20 (Estimated); Status verified 2014-03

CONDITIONS: Cystic Fibrosis; Chronic Obstructive Pulmonary Disease
Keywords: Respiratory health; Cystic Fibrosis; Chronic Obstructive Pulmonary Disease
MeSH Terms: conditions — Cystic Fibrosis; Pulmonary Disease, Chronic Obstructive

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Cross-Over Sequence 1 (Experimental): 85 μg GS-5737 in 2.8% saline or 2.8% saline alone (blinded)
  Interventions: Drug: GS-5737
- Cross-Over Sequence 2 (Experimental): 2.8% saline alone or 85 μg GS-5737 in 2.8% saline (blinded)
  Interventions: Drug: GS-5737

INTERVENTIONS:
Drug: GS-5737 — A single dose of GS-5737 in 2.8% saline

SUMMARY:
This is a randomized, double-blind, cross-over, vehicle-controlled study to determine whether GS-5737 in 2.8% saline accelerates mucociliary clearance (MCC) in healthy subjects, compared to vehicle of 2.8% saline alone.

ELIGIBILITY:
Inclusion Criteria:

* Body mass index (BMI) from ≥ 19 to ≤ 30 kg/m2
* Normal ECG, with no history or evidence of myocardial infarction, QT prolongation, or ventricular arrhythmias
* Normal (or abnormal but not clinically significant) blood pressure (BP) and heart rate(HR)
* History of lifetime smoking < 5 pack-years (ie, 1 pack per day x 1 year = 1 pack-year)and non-smokers of at least 60 days duration prior to Screening
* Negative screening tests for drugs of abuse (including alcohol)
* Hepatitis B (HBV) surface antigen negative
* Hepatitis C (HCV) antibody negative
* HIV-1, 2 antibody negative
* Male subjects who are sexually active must be willing to use highly effective contraception from the Baseline Visit through completion of the study and continuing for at least 90 days from the date of the last dose of study drug
* Male subjects must refrain from sperm donation from the Baseline Visit through completion of the study and continuing for at least 90 days from the date of the last dose of study drug
* Females of childbearing potential must have a negative serum pregnancy test
* Females of childbearing potential must agree to utilize protocol recommended highly effective contraception methods from Screening throughout the duration of study treatment and for 30 days following the last dose of study drug

Exclusion Criteria:

* Female subjects who are pregnant or lactating
* History of anaphylactic reaction to any drug
* Have previously participated in an investigational trial involving administration of any investigational compound within 30 days prior to the study drug dosing
* Presence or history of extrinsic allergy requiring treatment; hay fever is allowed unless it is active or has required treatment within the previous 2 months
* Have donated blood within 56 days of study dosing
* Presence or history of any pulmonary diseases (ie, asthma, emphysema, chronic bronchitis, chronic obstructive pulmonary disease (COPD), cystic fibrosis (CF), bronchiectasis, interstitial lung disease)
* Major surgery within 6 months of Screening
* Experienced symptoms of recent acute upper or lower respiratory tract infection requiring treatment within the 2 weeks prior to Screening
* Have had any radiation in the past year that would cause the subject exceed recommended limits by participating in this study protocol

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 7 (Actual)
Dates: Start 2012-10; Primary Completion 2013-06 (Actual); Study Completion 2013-06 (Actual)

PRIMARY OUTCOMES:
Area under the curve of MCC from Whole Lung Compartment | 4 weeks
  The primary endpoint of this study will be the calculated area under the curve of MCC from the whole lung compartment, assessed through 60 minutes post isotope dosing (AUC-60min), which will provide a description of the MCC curve.

SECONDARY OUTCOMES:
Area under the curve of MCC from Central and Peripheral Lung | 4 weeks or duration of study
  This outcome measure will be the calculated area under the cuve of MCC from the central and peripheral lung assessed through 60 minutes post isotope dosing (AUC60min).

OTHER OUTCOMES:
Safety and tolerability of GS-5737 | 4 weeks or duration of study
  Adverse events, airway reactivity, pulse oximetry, physical examination, and clinical laboratory test findings, urine and plasma potassium levels, 12-lead ECG abnormalities and interval measurements, and vital sign measurements will be used to assess this outcome measure.

CONTACTS AND LOCATIONS:
Overall Officials: Mark Bresnik, M.D., Study Director — Gilead Sciences
Locations (1):
- Investigational Site, Chapel Hill, North Carolina, United States